CLINICAL TRIAL: NCT05002335
Title: Clinical and Radiological Outcomes of Medacta Shoulder System (BE)
Status: Active, not recruiting | Type: Observational
Sponsor: Medacta International SA (Industry)
Responsible Party: Sponsor
Other Study IDs: P06.001.05
Record Dates: First submitted 2021-08-04; First posted 2021-08-12 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-06

CONDITIONS: Primary Osteoarthritis; Secondary Osteoarthritis; Rotator Cuff Tear Arthropathy; Rheumatoid Arthritis Shoulder; Avascular Necrosis; Fracture; Revision of Shoulder Arthroplasty
MeSH Terms: conditions — Rotator Cuff Tear Arthropathy; Osteonecrosis; Fractures, Bone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: Medacta Shoulder System — Performance of Total Shoulder Arthroplasty (anatomic/reverse) with Medacta Shoulder System

SUMMARY:
This is a post-market surveillance study on Medacta Shoulder System

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years
* Patient with one of the following diagnosis:

  1. Primary osteoarthritis
  2. Secondary osteoarthritis
  3. Cuff tear arthropathy; insufficient rotator cuff
  4. Acute fracture (<21d)
  5. Rheumatoid or inflammatory arthritis
  6. Avascular necrosis
  7. Other posttraumatic condition
  8. Revision of shoulder arthroplasty

Exclusion Criteria:

* Patients with malignant diseases (at the time of surgery)
* Patients with proven or suspect infections (at the time of surgery)
* Patients with functional deficits other than dysfunction of the shoulder (at the time of surgery)
* Patients with known incompatibility or allergy to products materials (at the time of surgery)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients requiring Total Shoulder Arthroplasty (anatomic/reverse) and who are suitable to receive Medacta Shoulder System will be proposed to take part to the current post-market surveillance study during their pre-operative visit.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-10-06 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Survival rate | 5 years
  Kaplan Meier method

SECONDARY OUTCOMES:
Clinical outcome; Constant and Murley score | 1, 2, and 5 years
  Constant & Murley Score: Its score ranges from 0 to 100 points, representing worst and best shoulder function, respectively. The pain experienced during normal activities of daily living was scored as: no pain = 15 points, mild = 10, moderate = 5 and severe = 0 points.
Functional outcome: Oxford Shoulder Score | 1, 2, and 5 years
  Oxford Shoulder Score: It contains 12 items, each with 5 potential answers. A mark between 1 (best/fewest symptoms) and 5 (worst/most severe) is awarded to correspond to the patient's symptoms. The combined total gives a minimum score of 12 and a maximum of 60. A higher score implies a greater degree of disability
Radiographic performance of the implants: Presence of radiolucencies | 3 months, 1, 2, and 5 years
  Presence of radiolucencies
Quality of life assesed by EQ-5D-5L score | 1, 2, and 5 years
  EQ-5D-5L score: The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
  The EQ VAS records the patient's self-rated health on a vertical visual analogue scale, where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'. The VAS can be used as a quantitative measure of health outcome that reflect the patient's own judgement.
Number of Intraoperative and postoperative Adverse events | intraop, 3 months, 1, 2, and 5 years
  Intraoperative and postoperative adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Bart Berghs, MD, Principal Investigator — AZ Sint-Jan (Brugge, Belgium)
Locations (3):
- Belgium (3):
  - AZ Sint-Jan, Bruges
  - AZ Sint-Lucas, Bruges
  - Clinique St-Luc Bouge, Namur

IPD SHARING:
Plan to Share IPD: No